CLINICAL TRIAL: NCT02873208
Title: A Phase 3, Multicenter Study to Assess the Long Term Safety and Tolerability of ALKS 3831 in Subjects With Schizophrenia
Brief Title: A Phase 3, Long-term Safety and Tolerability Study of ALKS 3831 in Adults With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK3831-A304
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
Keywords: Alkermes; ALKS 3831; Samidorphan; Schizophrenia; Safety
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALKS 3831 (Experimental): Oral tablet, daily dosing
  Interventions: Drug: ALKS 3831

INTERVENTIONS:
Drug: ALKS 3831 — Coated bilayer tablet containing 10 mg, 15 mg or 20 mg olanzapine and 10 mg samidorphan

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of ALKS 3831 in subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to use an acceptable method of contraception for the duration of the study
* Subject has completed the 24-week treatment period in the antecedent study, ALK3831-A303, within 7 days
* Additional criteria may apply

Exclusion Criteria:

* Subject is currently taking medications that are contraindicated with olanzapine use or exhibit drug-interaction potential with olanzapine
* Subject has a positive test for drugs of abuse at study entry
* Subject is pregnant, planning to become pregnant, or breastfeeding during the study
* Additional criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2016-08-07 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Principal Investigator — Alkermes, Inc.
Locations (42):
- United States (41):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Springdale, Arkansas
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Glendale, California
  - Alkermes Investigational Site, Lemon Grove, California
  - Alkermes Investigational Site, Long Beach, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, Redlands, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Temecula, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, Hollywood, Florida
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Augusta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Grand Rapids, Michigan
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, Creve Coeur, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Berlin, New Jersey
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigational Site, Brooklyn, New York
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, Rochester, New York
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Bellevue, Washington
- Alkermes Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects that had completed the 24-week treatment period of the antecedent study ALK3831-A303 within seven days prior to enrollment were eligible to be enrolled in the study.
Pre-assignment Details: One patient was enrolled and not dosed. A total of 265 patients were administered at least one dose of ALKS 3831 and included in the safety population.
Groups:
- ALKS 3831: All subjects assigned to ALKS 3831
  ALKS 3831: Coated bilayer tablet containing 10 mg, 15 mg or 20 mg olanzapine and 10 mg samidorphan
  Oral tablet, daily dosing
Period: Overall Study
Arm/Group | ALKS 3831
Started | 265
Completed | 167
Not Completed | 98
Not completed — Withdrawal by Subject | 36
Not completed — Lost to Follow-up | 22
Not completed — Adverse Event | 15
Not completed — Non-compliance with study drug | 12
Not completed — Protocol Violation | 8
Not completed — Pregnancy | 2
Not completed — Incarceration | 1
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | ALKS 3831
Number analyzed (Participants) | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 225
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 187
  White | 64
  More than one race | 6
  Unknown or Not Reported | 3
Height [Mean (Standard Deviation); unit: centimeters] | 173.24 (8.992)
Weight [Mean (Standard Deviation); unit: kilograms] | 80.64 (14.698)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 26.76 (3.756)
Body Mass Index (BMI) Group [Count of Participants; unit: Participants]
  Underweight (<18.5) | 1
  Normal (18.5 to <25) | 85
  Overweight (>=25 to <30) | 121
  Obese (>=30) | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Overall summary of treatment emergent adverse events during the treatment period
Time Frame: Up to 52 weeks
Population: Safety population was defined as all subjects who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 3831
Number analyzed (Participants) | 265
Participants
  Any Treatment Emergent Adverse Event (TEAE) | 161
  Mild Treatment Emergent Adverse Event (TEAE) | 93
  Moderate Treatment- Emergent Adverse Event (TEAE) | 61
  Severe Treatment- Emergent Adverse Event (TEAE) | 7
  Treatment- Emergent Adverse Event (TEAE)-Not Related | 82
  Treatment- Emergent Adverse Event (TEAE)-Related | 79
  Adverse Event Leading to Treatment Discontinuation | 15
  Any Serious Adverse Event (SAE) | 5
  Serious Adverse Event (SAE) -Not Related | 4
  Serious Adverse Event (SAE)-Related | 1
  Serious Adverse Event (SAE) leading to Death | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Groups:
- ALKS 3831: All subjects assigned to ALKS 3831 in ALKS 3831-A303 and ALKS 3831-A304
  ALKS 3831: Coated bilayer tablet containing 10 mg, 15 mg or 20 mg olanzapine and 10 mg samidorphan
  Oral tablet, daily dosing
Arm/Group | ALKS 3831
All-Cause Mortality (participants affected / at risk) | 0/265
Serious Adverse Events (participants affected / at risk) | 5/265
Other Adverse Events (participants affected / at risk) | 103/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 3831 (N=265)
Gastritis alcoholic (Gastrointestinal disorders) | 1
Schizophrenia (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 3831 (N=265)
Toothache (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Upper respiratory tract infection (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 10
Extra dose administered (Injury, poisoning and procedural complications) | 21
Weight decreased (Investigations) | 23
Weight increased (Investigations) | 16
Blood creatine phosphokinase increased (Investigations) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 9
Headache (Nervous system disorders) | 18
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT02873208/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02873208/SAP_001.pdf